CLINICAL TRIAL: NCT06411171
Title: Safety and Efficacy of Pembrolizumab in Combination With FLOT as a First-line Treatment in Patients With Gastroesophageal Junction Cancer: a Prospective Multicenter Randomized Controlled Trial
Brief Title: Safety and Efficacy of Pembrolizumab in Combination With FLOT About Gastroesophageal Junction Cancer:
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: xiaohua li (Other)
Responsible Party: Sponsor-Investigator, xiaohua li, associate chief physician, Xijing Hospital of Digestive Diseases
Organization: Xijing Hospital of Digestive Diseases (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KY20232301-F-1
Record Dates: First submitted 2024-05-07; First posted 2024-05-13 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Gastroesophageal Junction Cancer
MeSH Terms: interventions — pembrolizumab; Drug Therapy; Docetaxel; Oxaliplatin; Fluorouracil; Leucovorin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab plus chemotherapy (FLOT) (Experimental): Pembrolizumab plus chemotherapy (FLOT)
  Interventions: Drug: Pembrolizumab plus chemotherapy (FLOT)
- chemotherapy (FLOT) (Active Comparator): chemotherapy (FLOT)
  Interventions: Drug: Pembrolizumab plus chemotherapy (FLOT)

INTERVENTIONS:
Drug: Pembrolizumab plus chemotherapy (FLOT) — The experimental group was treated with pembrolizumab combined with FLOT, and the control group was treated with FLOT chemotherapy alone
  Other Names: docetaxel, oxaliplatin, fluorouracil, and leucovorin (the FLOT regimen)

SUMMARY:
At present, surgery is still the main treatment for gastroesophageal junction cancer. At the same time, multimodal comprehensive treatment such as chemotherapy and molecular targeted therapy can effectively alleviate pathological progression, facilitate R0 resection and improve the overall survival of patients.Pembrolizumab, as a PD-1 inhibitor, has been shown to have antitumor activity and a manageable safety profile in gastroesophageal junction cancer.Pembrolizumab combined with chemotherapy has become a research hotspot. However, to date, there is no clinical study related to gastroesophageal junction cancer. In this study, Pembrolizumab combined with FLOT was used as the first-line treatment for gastroesophageal junction cancer, aiming to explore the experience chemotherapy mode for gastroesophageal junction cancer.

DETAILED DESCRIPTION:
Gastric cancer, including gastroesophageal junction cancer, is the fifth most common cancer and the third leading cause of death in the world. Among them, although the incidence of distal gastric adenocarcinoma is decreasing, the incidence of gastroesophageal junction cancer is increasing. At present, surgery is still the main treatment for gastroesophageal junction cancer. At the same time, multi-mode comprehensive treatment such as chemotherapy and molecular targeted therapy can effectively alleviate pathological progression, facilitate R0 resection and improve the overall survival of patients. A large number of previous clinical trials on the combination of first-line chemotherapy and molecular targeted drugs in the treatment of gastric and gastroesophageal junction cancer have shown that only trastuzumab can improve the overall survival rate of Her-2 positive patients. In addition, despite various clinical chemotherapy regimens, the median survival time of gastric cancer and gastroesophageal junction cancer is not high. Therefore, the treatment mode of gastroesophageal junction cancer, especially for Her-2 negative patients, needs to be explored and improved.

In recent years, immune checkpoint inhibitors represented by programmed death receptor 1 (PD-1)/programmed death receptor ligand 1 (PD-L1) inhibitors have been applied to the treatment of a variety of solid tumors such as melanoma, non-small cell lung cancer, renal cell carcinoma, head and neck cancer, and urothelial cancer. It has become another important treatment strategy after surgery, chemotherapy, radiotherapy and targeted therapy. Studies have shown that PD-L1 is highly expressed in tumor cells and immune cells in gastric cancer and gastroesophageal junction cancer and plays a key role in tumor immune escape, therefore, the PD-1/ PD-L1 pathway will become an important target for effective intervention in gastroesophageal junction cancer. As a PD-1 inhibitor, Pembrolizumab has been shown to have anti-tumor activity and manageable safety in gastroesophageal junction cancer, and was approved by the US FDA in September 2017 for advanced PD-L1-positive gastric or gastroesophageal junction cancer . The phase Ⅱ KEYNOTE-059 trial used Pembrolizumab as a single agent in the third-line treatment of advanced gastric or gastroesophageal junction cancer, and the results showed that it had controllable safety in patients with PD-L1 positive, with obvious advantages in objective response rate (ORR) and median duration of response (DOR) [12]. Chemotherapy enhances tumor immune responses by enhancing tumor cell immunogenicity and sensitivity to immune killing, and the combination of chemotherapy and immune checkpoint inhibitors has been shown to improve overall survival in several cancer types. Therefore, PD-1/ PD-L1 immunosuppressant combined with chemotherapy has become a hot spot in the research of advanced gastric cancer or gastroesophageal junction cancer . The phase 3 KEYNOTE-062 trial compared Pembrolizumab plus chemotherapy (cisplatin plus 5-FU or capecitabine) with chemotherapy alone or Pembrolizumab alone in the first-line treatment of advanced gastric or gastroesophageal junction cancer. However, compared with chemotherapy alone, Pembrolizumab combined with chemotherapy could not significantly prolong the overall survival of patients, and the overall effect was not better than chemotherapy alone . In contrast, the phase III KEYNOTE-590 study, designed to compare the efficacy and safety of Pembrolizumab plus chemotherapy (cisplatin plus fluorouracil) versus chemotherapy alone as first-line treatment for advanced esophageal and Siwert type I gastroesophageal junction cancer, showed that Pembrolizumab combined with chemotherapy was significantly superior to chemotherapy alone . Neither the KEYNOTE-062 trial nor the KEYNOTE-590 trial analyzed a separate population of patients with gastroesophageal junction cancer, and there are some differences in response to drugs by tissue type. Therefore, The efficacy of Pembrolizumab plus chemotherapy in the only patient population with gastroesophageal junction cancer warrants further investigation.

ELIGIBILITY:
Inclusion Criteria:

* 1) aged from 18 to 75 years old, including 18 and 80 years old;

  2) histologically or cytologically confirmed locally advanced unresectable or metastatic gastric or GEJ adenocarcinoma;

  3) ECOG PS score 0 or 1;

  4) Known PD-L1 expression (assessed centrally using PD-L1 HC22C3)

  5) no previous treatment

  6) HER2-negative status

  7) normal hematological parameters: white blood cell count ≥4×109/L; Absolute neutrophil count ≥1.5×109/L; Platelet count ≥100×109/L; Blood red protein g/L;

  8) basically normal renal function: serum creatinine ≤1.5×ULN or creatinine clearance (CrCl)> 60 mL/min(using Cockcroft-Gault formula):

Female CrCl=(140-age)× weight (kg)× 0.85 / (72×Scr mg/dl)

Male CrCl=(140-age)× weight (kg)× 1.00 / (72×Scr mg/dl)

Liver function was basically normal: serum total bilirubin ≤1.5×ULN; Aspartate aminotransferase (AST) ≤2.5×ULN; Alanine aminotransferase (ALT) ≤2.5×ULN.

Female patients must have a negative urine pregnancy test before the start of the study (not applicable to patients with bilateral oophorectomy and/or hysterectomy or postmenopausal patients)

9) Provide written informed consent. Written informed consent was obtained.

Exclusion Criteria:

* 1) receiving anti-tumor therapy before enrollment, including but not limited to PD-1 inhibitors, CTLA-4 antibodies, EGFR monoclonal antibodies, EGFR-Tkis, and anti-angiogenic drugs;

  2) A history of autoimmune disease, including but not limited to: myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid syndrome-related vascular thrombosis, Wegener's granulomatosis, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, vasculitis, or glomerulonephritis. (Note: Patients with vitiligo, type I diabetes, or residual hypothyroidism due to autoimmune conditions (e.g., after Hashimoto's syndrome) requiring only hormone-replacement therapy, psoriasis requiring no systemic therapy, or if recurrence was not expected in the absence of an external trigger were allowed.) ;

  3) participated in other interventional clinical trials within 30 days before screening;

  4) Patients with a history of other malignant tumors (except cured basal cell carcinoma)

  5) with severe uncontrolled comorbidities (e.g., heart failure, diabetes mellitus, hypertension, liver failure, renal failure, thyroid disease, mental illness, etc.);

  6) known HIV infection or active viral hepatitis or tuberculosis;

  7) have a major surgical procedure or planned surgery within 30 days before the first dose of the trial drug;

  8) patients who are allergic to the drugs used in this regimen or their components;

  9) pregnant (confirmed by blood or urine HCG testing) or lactating women, or childbearing age subjects unwilling or unable to use effective contraception (for both male and female subjects) until at least 6 months after the last trial treatment;

  10) The investigator considers that it is not appropriate to participate in the study;

  11) unwilling to participate in the study or unable to sign an informed consent form

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
objective response rate | 3 year
  objective response rate

SECONDARY OUTCOMES:
duration of response | 1 year
  duration of response
disease control rate | 1 year
  disease control rate
time to response | 1 year
  time to response
overall surival | 5 year
  overall surival